CLINICAL TRIAL: NCT05108064
Title: Machine Learning Modeling the Risk of Refractory Pituitary Adenoma Using Radiomic and Pathomic Data
Brief Title: Radiomic and Pathomic Study of Pituitary Adenoma Using Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Clinical Professor, Huashan Hospital
Other Study IDs: KY2021-005
Record Dates: First submitted 2021-08-02; First posted 2021-11-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Artificial intelligence model — Results of artificial intelligence model will be compared with the gold standard

SUMMARY:
Refractory pituitary adenoma is characterized by invasive tumor growth, continuous growth and/or hormone hypersecretion in spite of standardized multi-modal treatment such as surgeries, medications or radiations. Quality of life or even lives are threatened by these tumors. According to the 2017 World Health Organization's new classification guideline of pituitary adenoma, patients have to suffer from symptoms or complications caused by these tumors, to bear a heavy financial burden, and to accept additional therapeutic side effects when the diagnosis of "refractory pituitary adenoma" is made. If refractory pituitary adenoma could be predicted at early stage, these patients would be able to have a more frequent clinical follow-up, receive multiple effective treatment as early as possible, or even be enrolled in clinical trials of investigational medications, so as to prevent or delay the recurrence or persistent of the tumor growth. Therefore, the unmet clinical need falls into an early prediction system for refractory pituitary adenomas, which could provide accurate guidance for subsequent treatment in the early stage. The investigators have constructed a pituitary adenoma database including clinical data, radiological images, pathological images and genetic information. The investigators are proposing a study using machine learning to extract features from these multi-dimensional, multi-omics data, which could be further used to train a prediction model for the risk of refractory pituitary adenoma. The proposed model would also be validated in another prospectively collected database. The established model would be able to identify potential medication targets and provide guidance for personalized therapy of refractory pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pituitary adenoma

Exclusion Criteria:

* Patients who were not able to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pituitary adenoma who were not able to sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The risk of refractory pituitary adenoma | 10 years
  Predicting the development of refractory pituitary adenoma after the first surgery

SECONDARY OUTCOMES:
Predicting Gamma Knife efficacy | 5 years
  Predicting endocrine remission after Gamma Knife surgery in Growth Hormone secreting pituitary adenoma
Predicting immunostaining | Two weeks after surgery
  Predicting immunostaining in patients with non-functioning pituitary adenoma using H&E stained images
Predicting recurrence | 10 years
  Predicting relapse or regrowth of a non-functioning pituitary adenoma after the first surgery
Predicting endocrinopathy | 10 years
  Predicting endocrinopathy which warrant replacement after pituitary adenoma resection
Predicting surgical difficulty and complications | Two weeks after surgery
  Predicting surgical difficulty and complications using pre-surgical radiomic features

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided